CLINICAL TRIAL: NCT05836909
Title: A Randomized, Double-blind, Placebo-controlled Trial of Using Red Yeast Rice, Phytosterol Esters and Lycopene in Combination for Regulating Lipid Metabolism of Guangzhou Individuals With Dyslipidemia
Brief Title: Regulation of Lipid Metabolism in Guangzhou Individuals With Dyslipidemia by Red Yeast Rice, Phytosterol Esters and Lycopene
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lili Yang (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor-Investigator, Lili Yang, head of Department of Nutrition, School of Public Health, Sun Yat-sen University, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Team Y
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Cholesterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swisse Plus cholesterol capsules (Experimental): (the main components are red yeast rice, phytosterol esters and lycopene)，the capsule is orally taken twice a day,two,tablets at a time 12 weeks
  Interventions: Dietary Supplement: Swisse plus cholesterol capsule
- placebo contral (Placebo Comparator): The placebo is an excipient and the colos, flavor, shape and weight are same with the Swisse plus cholesterol capsule
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Swisse plus cholesterol capsule — Swisse plus cholesterol capsule per day orally for 12 weeks
  Arms: Swisse Plus cholesterol capsules
Dietary Supplement: Placebo — Placebo
  Arms: placebo contral

SUMMARY:
The objective of this study is to evaluate the effect of using red yeast rice, phytosterol esters and lycopene in combination for 12 weeks on improving the glycolipid metabolism of Guangzhou individuals with dyslipidemia. Our hypothesis is that when compared with placebo, red yeast rice, phytosterol esters and lycopene together as supplements would lead to greater improvements in lipid metabolism (including lipid profiles and parameters ) in participants after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 30-50 years old.
2. Non-obese individuals: 18.5 ≤ BMI < 28.
3. Total cholesterol levels ranging from marginal increase to increase: 6.2> TC ≥ 5.2 mmol/L (200 mg/dL).

Exclusion Criteria:

1. Currently being pregnant or breast-feeding or planning to become pregnant.
2. Having severe complications of diabetes mellitus as well as any forms of cardiovascular diseases, tumor, liver diseases and kidney diseases.
3. History (past 3 months) of intake of lipid-lowering or anti-diabetic health care products.
4. Having hemorrhagic diathesis (high bleeding tendencies) or currently taking aspirin.
5. Unwilling/unable to draw blood due to physical/personal reasons.
6. History (past 1 month) of surgery.
7. History (past 1 month) of large amounts of oral or intravenous treatment of glucocorticoids (such as prednisone, methylprednisone, betamethasone, beclomethasone propionate, Dubossone, prednisone, hydrocodesone, dexamethasone).
8. History (past 2 weeks) of taking supplements containing red yeast rice, phytosterol ester or lycopene.
9. Unqualified outcomes of safety measures at baseline.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in levels of total cholesterol | 12 weeks
  At baseline, 4 weeks, 8 weeks and 12 weeks, bloods samples will be drawn and levels of total cholesterol will be determined in the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Lili Yang, Professor, Study Chair — Sun Yat-sen University
Locations (1):
- SunYat-senU, Guanzhou, Guangdong, China